CLINICAL TRIAL: NCT01604005
Title: PIT: A Phase III Randomised Trial of Prophylactic Irradiation of Tracts in Patients With Malignant Pleural Mesothelioma Following Invasive Chest Wall Intervention
Brief Title: PIT: Prophylactic Irradiation of Tracts in Patients With Malignant Pleural Mesothelioma
Acronym: PIT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: CI Decision:That once the last patient has reached 1 year follow-up, no further follow up needs to be completed on patients recruited in PIT"
Sponsor: Brynn Chappell (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Brynn Chappell, Clinical Trials Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08_DOG07_93; ISRCTN04240319 (Registry Identifier: ISRCTN); PB-PG-1010-23232 (Other Grant/Funding Number: NIHR Research for Patient Benefit)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; radiotherapy; prophylactic irradiation of tracts
MeSH Terms: conditions — Mesothelioma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIT Arm (Experimental)
  Interventions: Radiation: Prophylactic Irradiation of Tracts (PIT)
- No PIT Arm (No Intervention)

INTERVENTIONS:
Radiation: Prophylactic Irradiation of Tracts (PIT) — 21 Gy in 3 fractions
  Other Names: Radiation
  Arms: PIT Arm

SUMMARY:
The PIT (Prophylactic Irradiation of Tracts) trial will determine whether or not PIT radiotherapy is effective in preventing or delaying the onset of chest nodules in patients with Mesothelioma.

DETAILED DESCRIPTION:
Mesothelioma is a rare form of cancer affecting the protective lining that covers many of the body's internal organs. The most commonly affected areas are the lungs and internal chest wall. In the UK over 2300 patients are diagnosed with mesothelioma each year and the numbers are increasing.

As part of the diagnosis and treatment of mesothelioma, patients may undergo a procedure which involves inserting a thin tube into the chest wall enabling an internal examination and for any biopsies or samples of fluid to be taken. These procedures can result in the development of skin lumps or nodules along the tract created by inserting the tube. To try and reduce the risk of these nodules developing in the tract or at the site of the scar, radiotherapy can be given to the chest wall at the site of the tract after the procedure has been performed; this type of radiotherapy is known as prophylactic irradiation of tracts or PIT.

Although many hospitals already give patients this type of radiotherapy treatment to the chest wall we still do not know if the treatment works. This trial has been designed to answer the question about the effectiveness of PIT radiotherapy. If PIT is found to be effective in preventing or delaying the development of these skin nodules then it can be offered to all patients as part of their treatment. However, if we discover that PIT is not effective this will save patients from undergoing ineffective treatment and having to spend time making unnecessary extra visits to hospital

ELIGIBILITY:
Inclusion Criteria:

* Either sex, age ≥ 18 years
* Diagnosis of mesothelioma by multi-disciplinary team (MDT). All histological subtypes are eligible for the trial
* ECOG performance status 0-2 (Appendix C)
* Inoperable disease or operable disease in patients unsuitable for surgery as decided by a MDT
* Chest wall intervention with video-assisted thoracoscopy (VATS), open surgical biopsy (mini-thoracotomy), local anaesthetic thoracoscopy or chest drain
* Able to start radiotherapy within 42 days (6 weeks) of the most recent chest wall procedure
* Chest wall intervention scar visible at time of randomisation
* Radiotherapy target volume acceptable by the local radiotherapist
* Patients enrolled on other clinical trials could be considered after discussion with the chief investigators

Exclusion Criteria:

* Patients who underwent a thoracotomy (as large thoracotomy scars may not be adequately covered by this radiotherapy technique)
* Previous radiotherapy to the region of the chest wall intervention site
* Indwelling pleural catheter in-situ at the intervention site
* Patients currently receiving chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2012-07; Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of chest wall tract metastasis 6 months from randomisation | 6 months

SECONDARY OUTCOMES:
Time from randomisation to chest wall tract metastasis | Weeks
  Patients will be assessed at regular intervals approximately every 4 weeks by phone and at regular outpatient visits in the first year of follow up for signs of chest wall metastasis
Position of chest wall tract metastasis recurrence in relation to radiotherapy field in patients randomised to experimental arm (in field/out-of-field) | Weeks
  Patients will be assessed at regular intervals approximately every 4 weeks by phone and at regular outpatient visits in the first year of follow up for signs of chest wall metastasis
Acute and late skin radiotherapy toxicity | Weeks
  Patient will attend hospital at 6, 12, 26 and 52 weeks post randomisation where toxicity to PIT will be assessed.
  CTCAE v4.0 will be used
Pain from chest wall tract metastasis | Weeks
  Patients will be assessed at regular intervals approximately every 4 weeks by phone and at regular outpatient visits in the first year of follow for pain scoring using a Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, Study Chair — The Christie NHS Foundation Trust; Neil Bayman, Study Chair — The Christie NHS Foundation Trust
Locations (60):
- United Kingdom (60):
  - Tameside General Hospital, Ashton-under-Lyne
  - Basingstoke & North Hampshire Hospital, Basingstoke
  - Clatterbridge Cancer Centre, Bebington
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Royal Blackburn, Blackburn
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bolton Hospital, Bolton
  - Pilgrim Hospital, Boston
  - Bradford Royal Infirmary, Bradford
  - Queen's Hospital, Burton
  - Addenbrookes, Cambridge
  - Kent Oncology Centre, Canterbury
  - University Hospital of North Tees, Cleveland
  - University Hospital Coventry, Coventry
  - Leighton Hospital, Crewe
  - Royal Derby Hospitals, Derby
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Medway Maritime Hospital, Gillingham
  - The Royal Surrey County Hospital, Guildford
  - Princess Alexandra Hospital, Harlow
  - Harrogate District NHS Foundation Trust, Harrogate
  - Calderdale & Hudderfield NHS Trust, Huddersfield
  - Ipswich Hospital, Ipswich
  - St Mary's Hospital, Isle of Wight
  - Kidderminster General Hospital, Kidderminster
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - St James University Hospital, Leeds
  - University Hospital of Leicester, Leicester
  - United Lincolnshire Hospitals, Lincoln
  - North Middlesex Hospital, London
  - Macclesfield District General Hospital, Macclesfield
  - Maidstone Hospital, Kent Oncology Centre, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Wythenshawe Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Mount Vernon Cancer Centre, Middlesex
  - The Queen Elizabeth hospital, Norfolk
  - Northampton General Hospital, Northampton
  - Kings Mill Hospital, Nottingham
  - Nottingham University Hospitals, Nottingham
  - George Eliot Hospital, Nuneaton
  - Royal Oldham Hospital, Oldham
  - Peterborough City Hospital, Peterborough
  - Dorset Cancer Centre, Poole
  - Royal Preston Hospital, Preston
  - Glan Clwyd Hospital, Rhyl
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Sheffield Teaching Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - University Hospital of North Midlands, Stoke-on-Trent
  - Llandough Hospital, Vale of Glamorgan
  - Manor Hospital, Walsall
  - Warwick Hospital, Warwick
  - Wigan & Leigh NHS Foundation Trust, Wigan
  - New Cross Hospital, Wolverhampton
  - Alexandra Hospital, Worcestershire
  - York Teaching Hospital, York

REFERENCES:
- [Derived] Bayman N, Appel W, Ashcroft L, Baldwin DR, Bates A, Darlison L, Edwards JG, Ezhil V, Gilligan D, Hatton M, Jegannathen A, Mansy T, Peake MD, Pemberton L, Rintoul RC, Snee M, Ryder WD, Taylor P, Faivre-Finn C. Prophylactic Irradiation of Tracts in Patients With Malignant Pleural Mesothelioma: An Open-Label, Multicenter, Phase III Randomized Trial. J Clin Oncol. 2019 May 10;37(14):1200-1208. doi: 10.1200/JCO.18.01678. Epub 2019 Mar 28. PMID 30920878
- [Derived] Bayman N, Ardron D, Ashcroft L, Baldwin DR, Booton R, Darlison L, Edwards JG, Lang-Lazdunski L, Lester JF, Peake M, Rintoul RC, Snee M, Taylor P, Lunt C, Faivre-Finn C. Protocol for PIT: a phase III trial of prophylactic irradiation of tracts in patients with malignant pleural mesothelioma following invasive chest wall intervention. BMJ Open. 2016 Jan 27;6(1):e010589. doi: 10.1136/bmjopen-2015-010589. PMID 26817643
- See also: Christie NHS website — http://www.christie.nhs.uk/